CLINICAL TRIAL: NCT00050362
Title: Evaluation of a Long-Acting Local Anesthesia (Bupivacaine) and a Selective COX-2 Inhibitor (Rofecoxib) in Suppression of Central Sensitization
Brief Title: Rofecoxib and Bupivacaine to Prevent Pain After Third Molar (Wisdom Tooth) Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030055; 03-D-0055
Record Dates: First submitted 2002-12-04; First posted 2002-12-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Pain; Tooth Extraction
Keywords: Pain; NSAID; Oral Surgery; Hyperalgesia; Preemptive Analgesia
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — rofecoxib; Bupivacaine

INTERVENTIONS:
Drug: Rofecoxib and Bupivacaine

SUMMARY:
This study will evaluate the ability of the drugs rofecoxib and bupivacaine to prevent pain following third molar (wisdom tooth) extraction. Rofecoxib is approved to treat pain of arthritis and menstrual cramps. Bupivacaine is a local anesthetic similar to lidocaine, but longer acting.

Healthy normal volunteers between 16 and 35 years of age who are in general good health and require extraction of their two lower wisdom teeth may be eligible for this study.

Participants will have their two lower wisdom teeth extracted, and a biopsy (removal of a small piece of tissue) will be taken from the inside of the cheek around the area behind one of the extraction sites. Ninety minutes before surgery, patients will take a dose of either rofecoxib, or a placebo (a pill with no active ingredient) by mouth. Just before surgery, they will receive an injection of either lidocaine or bupivacaine to numb the mouth and a sedative called midazolam (Versed® (Registered Trademark)) through an arm vein to cause drowsiness. After surgery, a small piece of tubing will be placed into one of the two extraction sites. Samples will be collected from the tubing to measure chemicals involved in pain and inflammation.

Patients will remain in the clinic for up to 4 hours after surgery to monitor pain and drug side effects while the anesthetic wears off. During this time, they will complete pain questionnaires every 20 minutes. (Patients whose pain is unrelieved an hour after surgery may request and receive acetaminophen (Tylenol) and codeine.) The tubing then will be removed and they will be discharged with pain medicines (Tylenol, codeine and the study drug) and forms to record pain ratings. They will be given detailed instructions on how and when to take the medicines and how to record information in the pain diary.

Patients will return to the clinic 48 hours after surgery with the pain diary and pain relievers. At this visit, another biopsy will be taken under local anesthetic (lidocaine).

DETAILED DESCRIPTION:
Central sensitization refers to persistent post-injury changes in the central nervous system resulting in greater pain sensitivity. The concept of preemptive analgesia is defined as a treatment that prevents establishment of central sensitization by providing analgesic coverage during the perioperative period of surgery. Previous acute pain studies using the oral surgery model have shown that suppression of postoperative pain, not intra-operative nociceptive barrage, diminishes the development of sensitization at 24 to 48 hours post-surgery. During the intermediate postoperative period, the nociceptive input from both surgical insult and inflammation leads to central sensitization, yet their relative contributions have not been clearly evaluated. The proposed study is designed to evaluate the relative impact of surgical insult and the subsequent inflammation on postoperative pain. The relative contribution of each of these nociceptive processes provides a basis for postoperative pain management and the development of preemptive strategies.

All subjects (N = 136) will be healthy volunteers scheduled for third molar extractions. Using a double-blinded, randomized, parallel study design, subjects will be randomized into four groups. All patients will receive local anesthesia injections preoperatively (either 2% lidocaine or 0.5% bupivacaine) to manage surgical pain in conjunction with a preemptive medication (either 50 mg of rofecoxib or placebo) to control postoperative inflammation. The first dose of preemptive medication will be taken by mouth 90 minutes prior to conscious sedation and extractions, and later self-administered once a day for the next 48 hours. The analgesic effect of the drugs will be assessed in the clinic every 20 minutes for the first four hours after extractions, and then self-assessed at 24, and 48 hours after surgery using two pain intensity assessment instruments: category scale and visual analog scale (VAS). Microdialysis will be performed with sample collection concurrent with pain report over the immediate postoperative period of four hours. Two biopsies will be performed: preoperatively, and postoperatively at 48 hours. The combination regimen with bupivacaine and rofecoxib is predicted to maximally suppress the onset and intensity of postoperative dental pain to a greater extent than all other groups through a blockade of the nociceptive input from both surgery and inflammation. It is hypothesized that this preemptive treatment will maximally inhibit the development of central sensitization following tissue injury which manifests as hyperalgesia at later time points. It is also hypothesized that the administration of rofecoxib (a cyclooxygenase-2 selective anti-inflammatory medication) will reduce post-surgical pain experienced at later time points to a greater extent than suppression of the intra-operative nociceptive barrage alone (by bupivacaine), suggesting that suppression of inflammation plays a more pivotal role than attenuating nociception due to tissue injury in diminishing central sensitization.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female volunteers referred for third molar extraction willing to undergo 3 visits: 1 screening visit, 1 surgical appointment, and 1 follow-up research-related appointment.

Between the ages of 16-35 years (based upon eruption patterns and age-related complications associated with surgical extraction of third molars).

In general good health-American Society of Anesthesiologists (ASA) status I or II (healthy subjects based upon criteria for safe administration of out-patient conscious sedation).

Willing to undergo observation period for four hours postoperatively.

Willing to complete a 100 mm visual analog scale and a category scale every 20 minutes for the first 4 postoperative hours, and later at 24 and 48 hours.

Willing to have a microdialysis probe placed beneath the surgical flap over the first 4 hours post-surgery.

Willing to have a preoperative biopsy on the day of surgery and a postoperative biopsy at 48 hours.

Willing to return 48 hours post-operation to turn in completed pain diaries and for the postoperative biopsy.

Must have two lower partial (rating&eq;3) or fully impacted (rating&eq;4) wisdom teeth (mandibular third molars).

As assessed at the screening visit, the sum of the mandibular third molar surgical difficulty ratings must be between 6 to 8 in order to evaluate subjects experiencing similar pain levels.

EXCLUSION CRITERIA:

Allergy to aspirin, NSAIDs, or sulfites, amide anesthetics.

Pregnant or lactating females.

History of peptic ulcers and/or GI bleeding.

Chronic use of medications confounding the assessment of the inflammatory response or analgesia, for example, NSAIDS, COX-2 inhibitors, antihistamines, steroids, antidepressants.

Presence of a clinical sign suggestive of infection, inflammation or pre-existing pain.

Unusual surgical difficulty (determined from panoramic radiograph or during the actual surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136
Dates: Start 2002-12; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Woolf CJ. Evidence for a central component of post-injury pain hypersensitivity. Nature. 1983 Dec 15-21;306(5944):686-8. doi: 10.1038/306686a0. PMID 6656869
- [Background] Woolf CJ, Wall PD. Morphine-sensitive and morphine-insensitive actions of C-fibre input on the rat spinal cord. Neurosci Lett. 1986 Feb 28;64(2):221-5. doi: 10.1016/0304-3940(86)90104-7. PMID 3960401
- [Background] Cook AJ, Woolf CJ, Wall PD, McMahon SB. Dynamic receptive field plasticity in rat spinal cord dorsal horn following C-primary afferent input. Nature. 1987 Jan 8-14;325(7000):151-3. doi: 10.1038/325151a0. PMID 3808072